CLINICAL TRIAL: NCT04234893
Title: A Registry Study of Bingo Drug-Coated Balloon in Real World
Brief Title: Bingo Drug-Coated Balloon in Real World
Status: Completed | Type: Observational
Sponsor: Yinyi(Liaoning) Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: BEYOND Registry
Record Dates: First submitted 2020-01-06; First posted 2020-01-21 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Coronary Stenosis; Drug-coated Balloon; De Novo Stenosis; Coronary Artery Disease in Transplanted Heart Accelerated
Keywords: Coronary Stenosis; Percutaneous Coronary Intervention; Drug-coated Balloon; Drug eluting Balloon; Paclitaxel; De novo; Bifurcation; Coronary Artery Disease
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Drug-coated balloon: The Patients who treated with Bingo drug-coated balloon

SUMMARY:
The purpose is to observe and evaluate the safety and efficacy of Bingo drug-coated balloon in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older, regardless of gender;
2. Patients suitable for PCI with paclitaxel drug-coated balloon;
3. Patients able to understand the purpose of this study, provide an informed consent and cooperate with clinical follow-up.

Exclusion Criteria:

General exclusion criteria

1. Contraindications to PCI;
2. In-stent restenosis;
3. Life expectation less than 1 year;
4. Patients not suitable for enrollment considered by investigator.

Angiographic exclusion criteria:

1. Target lesion with the following conditions after pre-dilatation:

1. Residual stenosis larger than 30% ;
2. TIMI flow grade less than 3;
3. Type C-F dissection (NHLBI grade).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PCI with Bingo drug-coated balloon
Sampling Method: Probability Sample
Enrollment: 805 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 12 months
  a composite endpoint of cardiovascular death, myocardial infarction, clinical driven target lesion revascularization

SECONDARY OUTCOMES:
device success | immediately after the procedure
  study device successfully dilate in the lesion without using bail-out stent
lesion success | immediately after the procedure
  residual diameter stenosis ≤30% and the TIMI flow grade 3 of the target lesion
clinical success | immediately after the procedure， up to 7 days
  lesion success without in-hospital MACE
rate of Target lesion revascularization | 1, 6, 12 and 24 months
  repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Target lesion failure | 1, 6, 12 and 24 months
  a composite endpoint of cardiovascular death, target vessel myocardial infarction, clinical driven target lesion revascularization
Acute vessel closure | during the procedure and up to 24 hours
Target lesion thrombosis | immediately after the procedure， up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian-an Wang, MD, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China